CLINICAL TRIAL: NCT00877864
Title: Diabetes Exercise and Lifestyle Trial
Acronym: DEAL
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Dr. Ron Sigal, University of Calgary
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: DEAL- 22251; CHREB 22251
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; exercise; printed materials
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (6):
- High volume combined aerobic/resistance exercise (Active Comparator)
  Interventions: Behavioral: High volume combined aerobic/resistance exercise
- Low volume combined aerobic/resistance exercise (Active Comparator): Low volume combined aerobic/resistance exercise
  Interventions: Behavioral: Low volume combined aerobic/resistance exercise
- High volume combined A/R exercise, printouts, pedometers (Active Comparator): High volume combined aerobic/resistance exercise, printouts, pedometers
  Interventions: Behavioral: High volume combined A/R exercise, printouts, pedometers
- Low volume combined A/R exercise, printouts, pedometers (Active Comparator): Low volume combined aerobic/resistance exercise, printouts, pedometers
  Interventions: Behavioral: Low volume combined A/R exercise, printouts, pedometers
- Printed PA information, pedometers and step log group (Active Comparator): Printed physical activity information, pedometers and step log group
  Interventions: Behavioral: Printed PA information, pedometers and step log group
- Control (Placebo Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: High volume combined aerobic/resistance exercise — High volume combined aerobic/resistance exercise
  Arms: High volume combined aerobic/resistance exercise
Behavioral: Low volume combined aerobic/resistance exercise — Low volume combined aerobic/resistance exercise
  Arms: Low volume combined aerobic/resistance exercise
Behavioral: High volume combined A/R exercise, printouts, pedometers — High volume combined aerobic/resistance exercise, printouts, pedometers
  Arms: High volume combined A/R exercise, printouts, pedometers
Behavioral: Low volume combined A/R exercise, printouts, pedometers — Low volume combined aerobic/resistance exercise, printouts, pedometers
  Arms: Low volume combined A/R exercise, printouts, pedometers
Behavioral: Printed PA information, pedometers and step log group — Printed PA information, pedometers and step log group
  Arms: Printed PA information, pedometers and step log group
Behavioral: Control — No exercise program provided by the study
  Arms: Control

SUMMARY:
The objective of this study is to determine the effects of supervised combined aerobic and resistance training, and the effects of stage-matched written materials delivered by mail or internet, alone or in combination, on glycemic control as reflected in A1C (glycated hemoglobin).

DETAILED DESCRIPTION:
Background Rationale: Structured, supervised exercise programs involving aerobic exercise, resistance exercise or their combination resulted in significant improvements in glycemic control in type 2 diabetes. It has also been shown that programs which include a psychological/behavioral component in addition to diet and exercise have been most effective for long-term treatment of obesity in diabetes. The supervised exercise program has stronger evidence for improvement of metabolic control and cardiac risk, but its longer-term sustainability has not been demonstrated, and it is relatively costly. A stage-matched printed materials/pedometer intervention has been shown to increase physical activity over a longer period of time, and likely at a lower per-patient cost than the supervised exercise intervention, but with less evidence for improvement of metabolic control.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* A1c 0.700-0.099
* ability to read and write English
* signed ICF

Exclusion Criteria:

* participation in previous 6 months in exercise > 2 times per week for at least 20 min per session
* insulin therapy changes in medication for diabetes, BP or Lipids

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be A1c at the end of 6 months supervised exercise period. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ron Sigal, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada